CLINICAL TRIAL: NCT06447428
Title: One-Year Trajectory of Cognitive Changes in Patients With Late-life Depression in the Short Term: A Longitudinal Cohort Study
Brief Title: One-Year Trajectory of Cognitive Changes in Patients With Late-life Depression in the Short Term
Status: Recruiting | Type: Observational
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Zhu Ziping, Principal Investigator, Fujian Medical University
Other Study IDs: K2021-03-029
Record Dates: First submitted 2024-02-24; First posted 2024-06-07 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Late Life Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study was to investigate the one-year trajectory of cognitive change in elderly patients with depression, to explore the transfer characteristics and transfer rules of various states of cognitive impairment in patients, to predict the relevant risk factors of cognitive decline, and to find possible influencing factors affecting state change, so as to provide a theoretical basis and reference for subsequent targeted intervention research on geriatric depression.

DETAILED DESCRIPTION:
The 1-year prospective longitudinal study involved 400(prospective)subjects who met criteria for geriatric depression,the whole cognitive function was assessed by mini-mental state examination(MMSE),Montreal cognitive assessment scale-MOCA)and subjective cognitive decline scale(SCD-9).Cognitive function was monitored at 6 and 12 months.GAIN factors related to cognitive function(e.g.,age,gender,education,cognitive function,anxiety level,sleep,social support,resilience,social networks,etc.).By studying the longitudinal changes of cognitive function in the elderly patients with depression,a time-discrete and state-discrete multistate Markov model was constructed,namely,state 1(normal cognitive， NC),state 2(subjective cognitive decline， SCD),State 3(mild cognitive decline，MCI) and State 4(Alzheimer's disease，AD).In-depth analysis of some factors and indicators on the impact of the transfer between the states, the transfer between the states estimated probability.

ELIGIBILITY:
Inclusion Criteria:

1. meeting the criteria for major depression in the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5)
2. age at first onset ≥60 years
3. Informed consent

Exclusion Criteria:

1. Relevant past history affecting cognitive function: various types of stroke, traumatic brain injury, severe brain atrophy, mental abnormalities
2. Perennial alcohol addiction, or long-term use of various drugs that affect mental state
3. Survival time of malignant tumors and tumors
4. Patients with language, vision, and hearing impairments

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Elderly patients with depression who met the inclusion and exclusion criteria were selected from a number of nursing facilities, hospitals and communities
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Montreal cognitive assessment scale (MoCA) | 2023.6.1-2024.8.1
  The Changsha version of the MoCA questionnaire was used in this study, which included eight cognitive assessments of visuospatial and executive functions, naming, memory, attention, speech, abstraction, delayed recall, and orientation, with a total score of 30, with higher scores indicating better cognitive functioning.
Subjective cognitive decline questionnaire (SCD questionnaire 9, SCD-9) | 2023.6.1-2024.8.1
  The SCD-9 is mainly used to distinguish between normal people and SCD patients. The scale mainly consists of 2 dimensions, i.e., overall memory ability and time comparison (4 entries) and daily activity ability (5 entries), with a total of 9 entries, and the total scale score ranges from 0 to 9, with higher scores indicating a more severe degree of SCD.

SECONDARY OUTCOMES:
Activities of Daily Living (ADL) | 2023.6.1-2024.8.1
  The Activities of Daily Living (ADL) scale adopts a Liket four level rating. The evaluation results can be analyzed based on total score, dimension score, and individual score. A total score of 20 is considered completely normal, while a score above 20 indicates varying degrees of functional decline. A score of 1 for each item indicates normal functionality, while a score of 2-4 indicates decreased functionality.
general information | 2023.6.1-2024.8.1
  Using a self-made general information scale, such as age, gender, education level, and other basic personal information
Self Rating Anxiety Scale (SAS) | 2023.6.1-2024.8.1
  The Self Rating Anxiety Scale (SAS) has a total of 20 items, of which 5, 9, 13, 17, and 19 items are scored in reverse. The scale adopts a 1-4 level scoring method (1 point for no or very little time; 2 points for a small portion of time; 3 points for a considerable amount of time; 4 points for the vast majority or all of time). Individuals fill in the scale based on their own situation in the most recent week, multiply the calculated total score by 1.25, take an integer as the standard score, and use it as a statistical indicator. The higher the standard score, the more severe the anxiety level of the individual.
Social Support Rating Scale (SSRS) | 2023.6.1-2024.8.1
  The Social Support Rating Scale (SSRS) includes three dimensions: objective support, subjective support, and support utilization, with a total of 10 items: 1 point (none) to 4 points (full support). The higher the score in each dimension, the more support received.
Lubben Social Network Scale (LSNS-6) | 2023.6.1-2024.8.1
  The Lubben Social Network Scale (LSNS-6) is used to measure the structural characteristics of individual family and friend networks, as well as the supporting functions played by the network, in order to reflect the social network level of the respondents. It consists of two parts: the home network and the friend network, each with three items, totaling six items. Each entry has 5 options, with a score of 0-5 points and a total score of 0-30 points. The higher the score, the higher the level of social network, and<12 points indicates insufficient social network.
Pittsburgh Sleep Quality Index (PSQI) | 2023.6.1-2024.8.1
  The Pittsburgh Sleep Quality Index (PSQI) has a total of 19 items, divided into 7 components: subjective sleep quality, time to fall asleep, sleep time, sleep efficiency, sleep disorders, hypnotic drugs, and daytime function. The higher the total score, the worse the sleep quality.
Corner Davidson Resilience Scale (CDRISC) | 2023.6.1-2024.8.1
  The Corner Davidson Resilience Scale (CDRISC) consists of 10 items and uses the Likert 5-point scoring system. A score of 0-4 indicates "never", "rarely", "sometimes", "often", and "always", with higher scores indicating higher levels of psychological resilience.
Geriatric Depression Scale (GDS-15) | 2023.6.1-2024.8.1
  The Geriatric Depression Scale (GDS-15) is used to investigate the psychological feelings of patients in the past week. Result evaluation criteria: The total score range is 0-15 points, with higher scores indicating more severe depression. 1-5 points are subthreshold depression, 6-7 points are mild depression, 8-11 points are moderate depression, and 12-15 points are severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Ziping Zhu, Principal Investigator — Fujian Medical University
Locations (1):
- Fujian Medial University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Yes
Participant characteristics (e.g. age, gender, etc.), medical history (e.g. history of diabetes, hypertension, etc.), clinical outcomes (e.g. death), participation of patients at each stage, loss to follow-up rate
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2025.6-2026.6
Access Criteria: To obtain the data, you need to send an email address to the researcher himself